CLINICAL TRIAL: NCT00799760
Title: Evaluation of Combination Therapy With Oseltamivir and Zanamivir Versus Monotherapy in the Treatment of Virologically Confirmed Influenza in Primary Care a Randomises Double Blind Controlled Trial Study
Brief Title: Evaluation of Efficacity and Safety of Oseltamivir and Zanamivir
Acronym: BIVIR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Just Terminated for the end of the pandemia
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hoffmann-La Roche (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P060209; AOM 08209 (Other: French Ministry); 2008-004026-16 (EudraCT Number)
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2008-11

CONDITIONS: Gastric Influenza
Keywords: influenza A; neuraminidase inhibitor; oseltamivir; zanamivir; treatment outcome; resistance; mutation; combination therapy; monotherapy; pandemic; primary care; randomized controlled trials; antiviral agent
MeSH Terms: interventions — Oseltamivir; Zanamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): oral oseltamivir 75mg twice daily + zanamivir 10 mg inhaled by mouth twice daily during 5 days
  Interventions: Drug: oseltamivir + zanamivir
- 2 (Active Comparator): oral oseltamivir 75mg twice daily+ placebo inhaled by mouth twice daily during 5 days
  Interventions: Drug: oseltamivir + zanamivir's placebo
- 3 (Active Comparator): oral placebo twice daily + zanamivir 10 mg inhaled by mouth twice daily during 5 day
  Interventions: Drug: oseltamivir's placebo + zanamivir

INTERVENTIONS:
Drug: oseltamivir + zanamivir — oral oseltamivir 75mg twice daily + zanamivir 10 mg inhaled by mouth twice daily during 5 days
  Other Names: experimental Arm
  Arms: 1
Drug: oseltamivir + zanamivir's placebo — oral oseltamivir 75mg twice daily+ placebo inhaled by mouth twice daily during 5 day
  Other Names: Active comparator Arm
  Arms: 2
Drug: oseltamivir's placebo + zanamivir — oral placebo twice daily + zanamivir 10 mg inhaled by mouth twice daily during 5 day
  Other Names: active comparator arm
  Arms: 3

SUMMARY:
In order to prevent the high mortality due to an hypothetic pandemic caused by a newly emerging influenza A virus, antiviral drugs are seen as essential requirements for control of initial influenza outbreaks.Two antivirals are available for the treatment oseltamivir and zanamivir. Emergence of Oseltamivir resistance has been recently reported. . It appeared opportune to assess the efficacy and safety of biotherapy of neuraminidase inhibitors ,will be investigated by a randomized, placebo controlled, double blind study in France, during the next winter season . This study will be conducted in 300 centres of primary care with 900 adults with a virologically suspected influenza A infection. Individuals will be randomized to 1 of the 3 treatment groups: oseltamivir +zanamivir, or oseltamivir+placebo or placebo +zanamivir.The primary judgment criteria will be the proportion of patients with negative RT PCR negative in nasal secretions at Day 2.

DETAILED DESCRIPTION:
In the near future, a pandemic caused by a newly emerging influenza A virus has been predicted by the WHO. In order to prevent the high mortality due to the pandemic, antiviral drugs are seen as essential requirements for control of initial influenza outbreaks.

Zanamivir (GSK) and Oseltamivir (Roche) are stockpiled by the French government in the setting of pre-pandemic plan. In France, Zanamivir and Oseltamivir are both registered for the prophylactic and therapeutic use against influenza A.

Previous studies have shown that neuraminidase inhibitors (oseltamivir and zanamivir, based treatment) are associated with shorter illness duration and resulted in significant decrease of viral load in the nasal secretions.

In Winter season 2007-2008 the presence of oseltamivir-resistant viruses circulating in the community in several European countries is in marked contrast to the previous winter seasons, when oseltamivir resistance was detected in <1% of circulating strains from . Patients infected by viruses with neuraminidases carrying these mutations, didn't present unusual disease syndromes.

Although zanamivir and oseltamivir are both issued from the same class ,a combination of these two neuraminidase inhibitors could reduce the duration and severity of acute influenza and the incidence of secondary complications, reduce the spread of influenza, and the frequency of neuraminidase inhibitors mutations. An evaluation of the combination of oseltamivir and zanamivir versus zanamivir with placebo versus oseltamivir associated with placebo in the treatment of a virologically suspected influenza in primary care will be investigated in a randomised double blind placebo controlled trial study in France during the winter season 2008-2009.

Primary outcome measure:

Evaluate viral efficacy after 2 days of biotherapy oseltamivir and zanamivir versus zanamivir with placebo versus oseltamivir associated with placebo.

Patients and methods:

Randomised double blind, placebo controlled multicenter trial conducted during the influenza season 2008-2009 Arm 1: oral oseltamivir 75mg twice daily + zanamivir 10 mg inhaled by mouth twice daily during 5 days Arm 2: oral oseltamivir 75mg twice daily+ placebo inhaled by mouth twice daily during 5 days Arm 3: oral placebo twice daily + zanamivir 10 mg inhaled by mouth twice daily during 5 days.

Schedule:

D0: rapid test diagnostic for influenza A urine pregnancy test for women inclusion /randomisation initiation of treatment D2:nasal sample for influenza RNA RTPCR D5:End of treatment D7:medical evaluation (follow up evaluation) D14:nurse call (clinical evaluation)

ELIGIBILITY:
Inclusion Criteria:

* Influenza season declared
* Subjects aged>18 years presenting within 36h documented of onset influenza illness
* Who have fever >38°C
* who present at least on of the following respiratory symptoms( cough, sore throat, nasal symptoms)
* and one of the following constitutional symptoms(headache, myalgia, sweats and or chills or fatigue)
* positive rapid diagnostic test for influenza A
* who have giving written informed consent prior to enrollment
* Patient examined before the inclusion
* able to complete a questionnaire.

Exclusion Criteria:

* Influenza Vaccination in the 12 months prior the beginning of the study
* Patient unable to use diskhaler of Zanamivir
* Asthma, Chronic bronchitis,
* Woman with a positive urine pregnancy test
* Clearance of creatinine< 30 ml/min Chronic renal disease
* History of depression, psychiatric disorders
* oseltamivir or zanamivir hypersensibility
* patient treated by oseltamivir or zanamivir or amantadine 14 days before
* Non member of the social security or CMU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
RT-PCR for influenza A virus in nasal secretion | 2 days

SECONDARY OUTCOMES:
Time to resolution of influenzal illness Severity of illness | 14 days
Severity of illness | 14 Days
Adverse event (graded on a four -point scale:mild-moderate- severe-life threatening) | 14 days
Compliance to antiviral treatment | 14 days
Number of persons with influenza illness in households contact | 14 days
Evaluation of restricted activity (requirement for additional health car) | 14 days
Frequency of and need for antibiotic treatment of influenza (otitis media, bronchitis, sinusitis, and pneumonia ) | 14 days
Frequency of resistance to antiviral drugs | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Catherine LEPORT, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Centre Investigateur 155, Deûlémont, France

REFERENCES:
- [Result] Blanchon T, Mentre F, Charlois-Ou C, Dornic Q, Mosnier A, Bouscambert M, Carrat F, Duval X, Enouf V, Leport C; Bivir Study Group. Factors associated with clinical and virological response in patients treated with oseltamivir or zanamivir for influenza A during the 2008-2009 winter. Clin Microbiol Infect. 2013 Feb;19(2):196-203. doi: 10.1111/j.1469-0691.2011.03751.x. Epub 2012 Jan 20. PMID 22264308
- [Derived] Galimard JE, Chevret S, Curis E, Resche-Rigon M. Heckman imputation models for binary or continuous MNAR outcomes and MAR predictors. BMC Med Res Methodol. 2018 Aug 31;18(1):90. doi: 10.1186/s12874-018-0547-1. PMID 30170561
- [Derived] Flicoteaux R, Protopopescu C, Tibi A, Blanchon T, Werf SV, Duval X, Mosnier A, Charlois-Ou C, Lina B, Leport C, Chevret S. Factors associated with non-persistence to oral and inhaled antiviral therapies for seasonal influenza: a secondary analysis of a double-blind, multicentre, randomised clinical trial. BMJ Open. 2017 Jul 10;7(7):e014546. doi: 10.1136/bmjopen-2016-014546. PMID 28698321
- [Derived] Duval X, van der Werf S, Blanchon T, Mosnier A, Bouscambert-Duchamp M, Tibi A, Enouf V, Charlois-Ou C, Vincent C, Andreoletti L, Tubach F, Lina B, Mentre F, Leport C; Bivir Study Group. Efficacy of oseltamivir-zanamivir combination compared to each monotherapy for seasonal influenza: a randomized placebo-controlled trial. PLoS Med. 2010 Nov 2;7(11):e1000362. doi: 10.1371/journal.pmed.1000362. PMID 21072246